CLINICAL TRIAL: NCT05868473
Title: Effectiveness Of Mobilization With Movement And Kinesotaping In The Female Patients Of Knee Osteoarthritis To Improve Pain And Functional Mobility: A Randomized Controlled Trial
Brief Title: Effectiveness Of MM & Kinesotaping In The Female Patients Of KO To Improve Pain & Functional Mobility RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/527
Record Dates: First submitted 2023-03-18; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization With Movement (Other): Mobilization With Movement for Female Of Knee Osteoarthritis To Improve Pain And Functional Mobility
  Interventions: Diagnostic Test: Mobilization With Movement
- Kinesotaping (Experimental): Kinesotaping for Female Of Knee Osteoarthritis To Improve Pain And Functional Mobility
  Interventions: Diagnostic Test: Kinesotaping

INTERVENTIONS:
Diagnostic Test: Mobilization With Movement — Mobilization With Movement Female Of Knee Osteoarthritis To Improve Pain And Functional Mobility
  Arms: Mobilization With Movement
Diagnostic Test: Kinesotaping — Kinesotaping Female Of Knee Osteoarthritis To Improve Pain And Functional Mobility
  Arms: Kinesotaping

SUMMARY:
to find out the Effectiveness Of Mobilization With Movement And Kinesotaping In The Female Patients Of Knee Osteoarthritis To Improve Pain And Functional Mobility

ELIGIBILITY:
Inclusion Criteria:

* · Female patients of age ranging from age above 50 years suffering from knee Osteoarthritis will be included

Exclusion Criteria:

* · Patients suffering from any type of Cancer effecting area at which treatment will be applied.

  * Patients having joint replacement or knee disease effecting the performance.
  * Having skin allergies to taping.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
KOOS | 6 Months
  42 itens Questioner for Knee injury and Osteoarthritis Outcome Score
Li Scale | 6 Months
  Lequesne Index is an11-item questionnaire designed to obtain information of a subjective nature,

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No